CLINICAL TRIAL: NCT01721525
Title: Phase I Study of Induction Chemotherapy With Afatinib, Ribavirin, and Weekly Carboplatin/Paclitaxel for Stage IVA/IVB HPV Associated Oropharynx Squamous Cell Cancer (OPSCC)
Brief Title: Induction Chemotherapy With Afatinib, Ribavirin, and Weekly Carboplatin/Paclitaxel for Stage IVA/IVB HPV Associated Oropharynx Squamous Cell Cancer (OPSCC)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Comprehensive Cancer Network (Network); Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-150
Record Dates: First submitted 2012-11-01; First posted 2012-11-05 (Estimated); Last update posted 2017-10-25 (Actual); Status verified 2017-10

CONDITIONS: Head and Neck Cancer; Squamous Cell Cancer
Keywords: BIBW2992 (AFATINIB); CARBOPLATIN; RIBAVIRIN-ICN (VIRAZOLE); TAXOL (PACLITAXEL); OROPHARYNX; HPV associated; 12-150
MeSH Terms: conditions — Head and Neck Neoplasms; Neoplasms, Squamous Cell | interventions — Afatinib; Ribavirin; Paclitaxel; Jogging

ARMS (1):
- afatinib, ribavirin, and weekly carboplatin/paclitaxel (Experimental): This will be a single institution phase I study with an expansion cohort. Up to 2 dose levels of daily afatinib will be studied: 30 mg/day and 40 mg/day. The doses of ribavirin, carboplatin, and paclitaxel are fixed. A standard 3 + 3 phase I dose escalation design will be used.
  Interventions: Drug: Afatinib, Ribavirin, and weekly carboplatin/paclitaxel

INTERVENTIONS:
Drug: Afatinib, Ribavirin, and weekly carboplatin/paclitaxel — Patients will receive oral daily afatinib (days 1 - 21, per dose escalation scheme) plus daily oral ribavirin (days 1- 21) and paclitaxel (80 mg/m2 intravenously, days 1 and 8) + carboplatin (AUC 1.5 intravenously, days 1 and 8) of a 21-day cycle. Ribavirin will be administered according to standard weight-based dosing for this drug (1). Subjects ≤75 kg receive Ribavirin 400 mg PO qAM and 600 mg PO qPM (= 1000 mg/day). Subjects > 75 kg receive Ribavirin 600 mg PO BID (=1200 mg/day). During the Dose Escalation portion of the study (Part 1), research bloodwork for pharmacokinetics is performed on days 1 and 8 of Cycle 1 only.
  Other Names: During the Expansion Cohort (Part 2), there is a two week run in of afatinib +; ribavirin. The Expansion Cohort begins with a Run-In period of approximately; 14 days, in which patients receive only afatinib + ribavirin. On Day -14; (Start of the of the Run-In), patients begin afatinib once daily (at 40 mg/daily the dose; established in Part 1) and ribavirin twice daily according to standard; weight-based dosing. Both afatinib and ribavirin are self-administered each; day during the Run-In period.

SUMMARY:
This study seeks to develop a new induction chemotherapy regimen which is a combination of two pill drugs taken by mouth and two drugs given by vein. This is a phase I study, which means that the primary goal is to establish the recommended dose of an investigational drug when added to chemotherapy. The researchers wish to evaluate the effects, good and bad, of the investigational drug.

ELIGIBILITY:
Inclusion Criteria:

* Department of Pathology at MSKCC confirmation of diagnosis of oropharynx squamous cell cancer, stage IVA/IVB, that is HPV associated.

Evidence of HPV can be p16 immunohistochemistry and/or HPV in situ hybridization positive test result on tumor tissue, either at MSKCC or other CLIA-approved lab.

* Age ≥ 18 years of age
* Karnofsky Performance Status ≥ 80
* Adequate organ function, as follows:

Adequate bone marrow reserve: absolute neutrophil count (ANC) ≥ 1.5 X 109/L, platelets ≥ 160 X 109/L, hemoglobin ≥ 12 g/dL Hepatic: total bilirubin within normal limits (≤ 1.0 mg/dL); alkaline phosphatase (AP), aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 1.5 X ULN (upper limit of normal) Renal: Serum creatinine ≤ 1.3 mg/dL. Patients with serum creatinine > 1.3 mg/dL may be eligible if creatinine clearance (CrCl) ≥ 55 mL/min based on the standard Cockroft and Gault formula.

* Patients of childbearing potential must have a negative serum pregnancy test within 14 days of treatment. Patients must agree to use a reliable method of birth control during and for 6 months following the last dose of study drug.
* Ability to swallow oral medication.
* Expansion Cohort only: At least one unstained slide from pre-treatment diagnostic biopsy or fine needle aspirate must be available for correlative immunohistochemistry study.

Exclusion Criteria:

* Prior chemotherapy or radiation for tonsillar or base of tongue squamous cell cancer
* History of hemolytic anemia or thalassemia
* Active infection or serious underlying medical condition that would impair the patient's ability to receive protocol treatment.
* Current therapeutic anticoagulation with Coumadin (warfarin)
* Current or prior treatment with ribavirin
* Known active Hepatitis B or C
* Any prior documented history of transient ischemic attack (TIA) or cerebrovascular accident (CVA)
* New York Heart Association (NYHA) Grade II or greater congestive heart failure
* Clinically significant peripheral vascular disease
* Inability to discontinue any of the following potent P-gp inhibitors (cyclosporine, erythromycin, ketoconazole, itraconazole, quinidine, phenobarbital salt with quinidine, ritonavir, valspodar, verapamil) or inducers (St John's wort, rifampicin).
* Known pre-existing interstitial lung disease.
* Presence of poorly controlled gastrointestinal disorders that could affect the absorption of the trial drug (e.g. Crohn's disease, ulcerative colitis, malabsorption, or CTC grade ≥2 diarrhea of any etiology) based on treating physician assessment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-11 (Actual); Primary Completion 2017-10-16 (Actual); Study Completion 2017-10-16 (Actual)

PRIMARY OUTCOMES:
maximum tolerated dose (For Dose Escalation Portion of the study) | 1 year
  of daily oral afatinib administered with standard daily weight based ribavirin and intravenous carboplatin and paclitaxel, Up to 2 dose levels of daily afatinib will be studied: 30 mg/day and 40 mg/day. The doses of ribavirin, carboplatin, and paclitaxel are fixed. A standard 3 + 3 phase I dose escalation design will be used.
expression of PTPN13 (For Expansion Cohort only) | 1 year
  To determine if a two week run-in with afatinib and ribavirin results in increased expression of PTPN13, as determined by IHC in pre and post treatment biopsies.

SECONDARY OUTCOMES:
safety and tolerability (toxicity) | 1 year
  Adverse events (AEs) will be assessed according to NCI common toxicity criteria (CTC) version 4.0. Dose Limiting Toxicity (DLT) include all toxicities of grade 3 or higher felt to be possibly, probably, or definitely related to study drug.
objective response rate | 1 year
  Response and progression will be evaluated in this study using modified international criteria proposed by the revised Response Evaluation Criteria in Solid Tumors (RECIST) guideline (version 1.1) (51). Changes in the largest diameter (unidimensional measurement) of the tumor lesions and the shortest diameter in the case of malignant lymph nodes are used in the RECIST criteria.
pharmacokinetics | 1 year
  PK measurements will be collected from patients in the dose excalation cohort during the first cycle of therapy. The area under the curve (AUC0→∞), half-life (t½), and maximum concentration (Cmax) for afatinib will be determined by noncompartmental analysis.

CONTACTS AND LOCATIONS:
Overall Officials: David Pfister, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (2):
- United States (2):
  - Memorial Sloan Kettering Cancer Center at Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Cancer Center, New York, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/